CLINICAL TRIAL: NCT01199887
Title: A Phase One, Open Label, Multi-Dose Study to Evaluate the Safety, Tolerability, and Biologic Effects of Three Doses of IW001 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Trial Of IW001 in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneWorks (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IW001-01
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: safety, biologic effects, IPF, autoimmune
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IW001 (Experimental): Three dose cohorts, 0.1 mg, 0.5 mg, 1.0 mg
  Interventions: Drug: IW001

INTERVENTIONS:
Drug: IW001 — IW001, 0.1 mg, 0.5 mg, 1.0 mg PO daily for 24 weeks.

SUMMARY:
This is an open label, Phase One, multicenter study, designed to evaluate the safety, tolerability, to explore the biologic effects, and to explore the clinical effects of the following doses of IW001: 0.1mg/day, 0.5 mg/day, and 1.0 mg/day, when administered once a day orally for 24 weeks in patients with IPF.

DETAILED DESCRIPTION:
IW001 is a therapeutic designed to treat anti-Col (V)-mediated autoimmune diseases via oral tolerance. With the identification of the specific antigen involved in the autoimmune disease process in IPF, IW001 induced oral tolerance may be an effective treatment. IW001 is taken orally, introduced into the mucosal immune system at the Peyer's Patches in the distal small intestine, where antigen-presenting cells present the antigen to regulatory T cells (Tregs). These antigen-specific Tregs enter the blood stream and traffic to areas where the specific antigen has generated an autoimmune response. Thus, IW001 may produce selective suppression of immune responses against Col (V).

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following to be included in the study:

  1. Diagnosis of IPF (ATS criteria) prior to the Baseline visit.
  2. Forced Vital Capacity (FVC) ≥ 50% of predicted.
  3. Lung Diffusion Capacity (DLCO) ≥ 35% of predicted.
  4. Ages 35-75 years inclusive.
  5. Positive for anti-Col (V) antibodies.
  6. White blood cell count (WBC) ≥ 2500 mm3.
  7. Hematocrit ≥ 25% and ≤ 59%.
  8. Platelets ≥ 100,000 mm3.
  9. Creatinine ≤ 1.5x Upper Limits of Normal (ULN).
  10. Bilirubin ≤ 1.5x ULN.
  11. Aspartate aminotransferase (AST, SGOT) ≤ 1.5x ULN.
  12. Females of child-bearing potential (defined as less than one year post-menopausal or not surgically sterile) must be using an acceptable method of birth control or practicing abstinence from the time consent is signed until 30 days after treatment discontinuation. If sexually active, female patients must use a double barrier method of birth control, such as a condom and spermicidal. Patient must have a negative pregnancy test at the Screening and Baseline visits.
  13. Willing and able to provide adequate written informed consent.

      Exclusion Criteria:
* Patients will be excluded from the study for any of the following:

  1. Concurrent use of systemic corticosteroids or immunosuppressives within 30 days of the Baseline visit.
  2. Chronic NSAID use (limited, i.e., up to 72 hours continuous use of NSAIDs will be permitted during the study), (see Section 9, concomitant medications).
  3. N-acetyl cysteine (NAC) use within 14 days of the Baseline visit.
  4. Any disease, condition or surgery (e.g. inflammatory bowel disease, surgical resection) that may cause malabsorption of IW001.
  5. Known or suspected allergy to bovine products.
  6. Concurrent or prior use of any experimental medication within 30 days of the Baseline visit.
  7. History of smoking within three months prior to the Baseline visit.
  8. Known Hepatitis C or Human Immunodeficiency Virus (HIV) infections.
  9. Evidence of active infection at the Baseline visit.
  10. History of unstable or deteriorating cardiac disease.
  11. Myocardial infarction, coronary artery bypass, or angioplasty within 6 months of the Baseline visit.
  12. Unstable angina pectoris or congestive heart failure requiring hospitalization within 6 months of the Baseline visit.
  13. Uncontrolled arrhythmia.
  14. Patient has a history of illicit drug or alcohol abuse in the past year or current evidence of such abuse or addiction in the opinion of the Investigator.
  15. Patient has positive findings on urine drug screen.
  16. Any other clinically significant illness, that, in the opinion of the Investigator, might put the patient at risk of harm during the study or might adversely affect the interpretation of the study data.
  17. Females who are pregnant and/or lactating.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of three doses of IW001 (0.1 mg/day, 0.5 mg/day, and 1.0 mg/day orally) in patients with IPF patients over a 24 week treatment period. | Monthly during the 24 week treatment period.

SECONDARY OUTCOMES:
To explore the biologic effects of IW001 on T-cell and B-cell reactivity. To explore relationships between Col V reactivity and clinical measures of lung function in patients with IPF. | Monthly during the 24 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Chew, MD, Study Director — ImmuneWorks, Medical Consultant
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - IUPUI, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Newark Beth Israel Hospital, Newark, New Jersey
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Background] American Thoracic Society. Idiopathic pulmonary fibrosis: diagnosis and treatment. International consensus statement. American Thoracic Society (ATS), and the European Respiratory Society (ERS). Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):646-64. doi: 10.1164/ajrccm.161.2.ats3-00. No abstract available. PMID 10673212
- [Background] Raghu G, Weycker D, Edelsberg J, Bradford WZ, Oster G. Incidence and prevalence of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2006 Oct 1;174(7):810-6. doi: 10.1164/rccm.200602-163OC. Epub 2006 Jun 29. PMID 16809633
- [Background] Martinez FJ, Safrin S, Weycker D, Starko KM, Bradford WZ, King TE Jr, Flaherty KR, Schwartz DA, Noble PW, Raghu G, Brown KK; IPF Study Group. The clinical course of patients with idiopathic pulmonary fibrosis. Ann Intern Med. 2005 Jun 21;142(12 Pt 1):963-7. doi: 10.7326/0003-4819-142-12_part_1-200506210-00005. PMID 15968010
- [Background] Walter N, Collard HR, King TE Jr. Current perspectives on the treatment of idiopathic pulmonary fibrosis. Proc Am Thorac Soc. 2006 Jun;3(4):330-8. doi: 10.1513/pats.200602-016TK. PMID 16738197
- [Background] Trulock EP, Edwards LB, Taylor DO, Boucek MM, Keck BM, Hertz MI. Registry of the International Society for Heart and Lung Transplantation: twenty-second official adult lung and heart-lung transplant report--2005. J Heart Lung Transplant. 2005 Aug;24(8):956-67. doi: 10.1016/j.healun.2005.05.019. No abstract available. PMID 16102428
- [Background] Kim DS, Collard HR, King TE Jr. Classification and natural history of the idiopathic interstitial pneumonias. Proc Am Thorac Soc. 2006 Jun;3(4):285-92. doi: 10.1513/pats.200601-005TK. PMID 16738191
- [Background] Maher TM, Wells AU, Laurent GJ. Idiopathic pulmonary fibrosis: multiple causes and multiple mechanisms? Eur Respir J. 2007 Nov;30(5):835-9. doi: 10.1183/09031936.00069307. PMID 17978154
- [Background] Hunninghake GW, Schwarz MI. Does current knowledge explain the pathogenesis of idiopathic pulmonary fibrosis? A perspective. Proc Am Thorac Soc. 2007 Aug 15;4(5):449-52. doi: 10.1513/pats.200702-036MS. PMID 17684287
- [Background] Bobadilla JL, Love RB, Jankowska-Gan E, Xu Q, Haynes LD, Braun RK, Hayney MS, Munoz del Rio A, Meyer K, Greenspan DS, Torrealba J, Heidler KM, Cummings OW, Iwata T, Brand D, Presson R, Burlingham WJ, Wilkes DS. Th-17, monokines, collagen type V, and primary graft dysfunction in lung transplantation. Am J Respir Crit Care Med. 2008 Mar 15;177(6):660-8. doi: 10.1164/rccm.200612-1901OC. Epub 2008 Jan 3. PMID 18174545
- [Background] Burlingham WJ, Love RB, Jankowska-Gan E, Haynes LD, Xu Q, Bobadilla JL, Meyer KC, Hayney MS, Braun RK, Greenspan DS, Gopalakrishnan B, Cai J, Brand DD, Yoshida S, Cummings OW, Wilkes DS. IL-17-dependent cellular immunity to collagen type V predisposes to obliterative bronchiolitis in human lung transplants. J Clin Invest. 2007 Nov;117(11):3498-506. doi: 10.1172/JCI28031. PMID 17965778
- [Background] Faria AM, Weiner HL. Oral tolerance. Immunol Rev. 2005 Aug;206:232-59. doi: 10.1111/j.0105-2896.2005.00280.x. PMID 16048553
- [Background] Whitacre CC, Song F, Wardrop RM 3rd, Campbell K, McClain M, Benson J, Guan Z, Gienapp I. Regulation of autoreactive T cell function by oral tolerance to self-antigens. Ann N Y Acad Sci. 2004 Dec;1029:172-9. doi: 10.1196/annals.1309.033. PMID 15681756
- [Background] Nussenblatt R. Orally and nasally induced tolerance studies in ocular inflammatory disease: guidance for future interventions. Ann N Y Acad Sci. 2004 Dec;1029:278-85. doi: 10.1196/annals.1309.058. PMID 15681765
- [Background] Artik S, Haarhuis K, Wu X, Begerow J, Gleichmann E. Tolerance to nickel: oral nickel administration induces a high frequency of anergic T cells with persistent suppressor activity. J Immunol. 2001 Dec 15;167(12):6794-803. doi: 10.4049/jimmunol.167.12.6794. PMID 11739495
- [Background] Barnett ML, Kremer JM, St Clair EW, Clegg DO, Furst D, Weisman M, Fletcher MJ, Chasan-Taber S, Finger E, Morales A, Le CH, Trentham DE. Treatment of rheumatoid arthritis with oral type II collagen. Results of a multicenter, double-blind, placebo-controlled trial. Arthritis Rheum. 1998 Feb;41(2):290-7. doi: 10.1002/1529-0131(199802)41:23.0.CO;2-R. PMID 9485087
- [Background] McKown KM, Carbone LD, Bustillo J, Seyer JM, Kang AH, Postlethwaite AE. Induction of immune tolerance to human type I collagen in patients with systemic sclerosis by oral administration of bovine type I collagen. Arthritis Rheum. 2000 May;43(5):1054-61. doi: 10.1002/1529-0131(200005)43:53.0.CO;2-W. PMID 10817559
- [Background] Carbone LD, McKown K, Pugazhenthi M, Barrow KD, Warrington K, Somes G, Postlethwaite AE. Dosage effects of orally administered bovine type I collagen on immune function in patients with systemic sclerosis. Arthritis Rheum. 2004 Aug;50(8):2713-5. doi: 10.1002/art.20361. No abstract available. PMID 15334493
- [Background] Postlethwaite AE, Wong WK, Clements P, Chatterjee S, Fessler BJ, Kang AH, Korn J, Mayes M, Merkel PA, Molitor JA, Moreland L, Rothfield N, Simms RW, Smith EA, Spiera R, Steen V, Warrington K, White B, Wigley F, Furst DE. A multicenter, randomized, double-blind, placebo-controlled trial of oral type I collagen treatment in patients with diffuse cutaneous systemic sclerosis: I. oral type I collagen does not improve skin in all patients, but may improve skin in late-phase disease. Arthritis Rheum. 2008 Jun;58(6):1810-22. doi: 10.1002/art.23501. PMID 18512816
- [Background] Baccarani U, Adani GL, Montanaro D, Risaliti A, Lorenzin D, Avellini C, Tulissi P, Groppuzzo M, Curro G, Luvisetto F, Beltrami A, Bresadola V, Viale PL, Bresadola F. De novo malignancies after kidney and liver transplantations: experience on 582 consecutive cases. Transplant Proc. 2006 May;38(4):1135-7. doi: 10.1016/j.transproceed.2006.02.016. PMID 16757287
- [Background] Yasufuku K, Heidler KM, O'Donnell PW, Smith GN Jr, Cummings OW, Foresman BH, Fujisawa T, Wilkes DS. Oral tolerance induction by type V collagen downregulates lung allograft rejection. Am J Respir Cell Mol Biol. 2001 Jul;25(1):26-34. doi: 10.1165/ajrcmb.25.1.4431. PMID 11472972
- [Background] Mizobuchi T, Yasufuku K, Zheng Y, Haque MA, Heidler KM, Woods K, Smith GN Jr, Cummings OW, Fujisawa T, Blum JS, Wilkes DS. Differential expression of Smad7 transcripts identifies the CD4+CD45RChigh regulatory T cells that mediate type V collagen-induced tolerance to lung allografts. J Immunol. 2003 Aug 1;171(3):1140-7. doi: 10.4049/jimmunol.171.3.1140. PMID 12874199